CLINICAL TRIAL: NCT01822301
Title: Structural Fat Grafting for Craniofacial Trauma: Repeat Fat Grafting Injection-5 Subject Cohort
Acronym: BTIPlusUp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, J. Peter Rubin, MD, Founding Chair Department of Plastic Surgery Professor of Surgery at the University of Pittsburgh School of Medicine, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO12100585
Record Dates: First submitted 2013-03-19; First posted 2013-04-02 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Facial Injuries; Adipose Tissue
Keywords: Craniomaxillofacial (CMF) Battle-injured (BI); Facial Trauma; Fat Grafts; Autogenous Fat Transfers (AFT); Wounded warriors
MeSH Terms: conditions — Facial Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Repeat Facial fat grafting (Experimental)
  Interventions: Procedure: Repeat Fat grafting

INTERVENTIONS:
Procedure: Repeat Fat grafting — Fat grafting is a minimally invasive clinical procedure that has been widely used by plastic surgeons within reconstructive surgery for many years. Fat grafting is considered a standard of care procedure in plastic surgery. In brief, fat tissue to be used for grafting is harvested (usually from abdomen or thighs) with a small liposuction cannula in the operating room. The fat tissue is then sterilely centrifuged and allowed to decant before separating the fluid and oil layers from the fat tissue fraction. The aspirated fat is then loaded into 1cc syringes and injected into the facial deformity using specialized injection cannulas. In this study, we will treat 5 subjects from protocol (IRB # PRO09060101) with an additional fat graft treatment to assess whether this will increase fat graft retention over time. Additionally, data from our current study assessing volume retention after fat grafting for facial deformities (IRB # PRO09060101) with be used for comparison.

SUMMARY:
Fat grafting represents a technique with great potential to improve outcomes in minimally invasive facial reconstruction. Fat grafting has already been demonstrated as a safe and minimally invasive technique over decades of widespread practice in plastic surgery. In our current study of fat grafting for facial deformities (IRB# PRO09060101), we have treated 9 subjects without adverse event and all have had a significant improvement. Since all methods of treatment and evaluation are the same in this study, we will be able to use the data in our prior study as additional control data.

We hypothesize that repeating the fat grafting in subjects with previous facial fat grafts will enable successful restoration of tissue volume and craniofacial form. Additionally, we hypothesize that the results will be durable and subject quality of life improved.

Five (5) subjects (who were previously enrolled into IRB# PRO09060101) will be enrolled to this single center University of Pittsburgh site research study.

DETAILED DESCRIPTION:
Facial trauma injuries, especially those sustained in military combat and severe automobile crashes, are characterized by destruction of bone and soft tissue anatomy. While the bony skeleton can often be reconstructed, the overlying soft tissue is difficult to restore.

Importantly, it is the structure of the soft tissue that imparts the normal human form, and adequate reconstruction of soft tissue defects allows trauma victims to reintegrate into society. Accepted procedures for soft tissue reconstruction of the face involve tissue flap reconstruction procedures and autologous fat grafting. Tissue flap operations are extensive, often including microvascular surgery, and do not precisely correct the deformities. Fat grafting is a less invasive technique that allows for more precise shaping of the reconstructed tissues. However, autologous fat grafts may undergo resorption that can affect the appearance of the reconstruction over time. The degree of change in appearance after fat grafting has not been well studied for facial trauma patients.

We hypothesize that subjects who have successfully completed participation in the study (PRO09060101) and experienced graft resorbtion will have improved outcomes with an additional fat graft treatment. We anticipate that additional fat graft treatment will fully restore the facial features and overcome fat loss from the initial fat graft treatment. Additionally, we hypothesize that the cellular properties of the fat precursor cells (preadipocytes) may correlate with fat graft retention

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older and able to provide informed consent
2. Have suffered injury resulting in craniofacial volume defects which could be treated with a graft volume of between 5 and 150 cc of lipoaspirate
3. Be at least 3 months post-injury or post-surgery (from trauma procedures) so that acute edema is resolved
4. Volume defects are covered by intact skin and do not communicate with oral cavity or sinuses
5. The three dimensional geometry of the volume defects would allow for treatment with lipoaspirate injection that in a manner that at least two distinct treated areas could be discerned on gross examination and radiographically (e.g. treated regions are on opposite sides of the face, on lower face versus upper face, or separated by a bony landmark such as zygoma. This would include the ability to treat an uninjured contralateral region with lipaspirate in order to obtain symmetry.
6. Willing and able to comply with follow up examinations, including radiographic studies
7. Have completed participation in IRB# PRO09060101.

Exclusion Criteria:

1. Age less than 18 years
2. Inability to provide informed consent
3. Craniofacial defects intended for treatment have open wounds or communicate with oral cavity or sinus (note: presence of such a defect in the setting of another defect(s) that meets treatment criteria will not exclude the patient from participating).
4. Active infection anywhere in the body
5. Diagnosed with cancer within the last 12 months and /or presently receiving chemotherapy or radiation treatment
6. Known coagulopathy
7. Systemic disease that would render the fat harvest and injection procedure, along with associated anesthesia, unsafe to the patient.
8. Pregnancy
9. Subjects with Schizophrenia, Bipolar Disorder. (Subjects who are found to be stable on medication and receive psychiatric clearance could be eligible for study participation per the Physician's discretion.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Rubin, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Unversity of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
It is the Principal Investigator's intention to make stored samples and subject de-identified information available to secondary investigators after all research study testing has been completed. These stored samples and associated subject information will not include subject identifiers.

REFERENCES:
- [Background] Moseley TA, Zhu M, Hedrick MH. Adipose-derived stem and progenitor cells as fillers in plastic and reconstructive surgery. Plast Reconstr Surg. 2006 Sep;118(3 Suppl):121S-128S. doi: 10.1097/01.prs.0000234609.74811.2e. PMID 16936551
- [Background] Cardenas JC, Carvajal J. Refinement of rhinoplasty with lipoinjection. Aesthetic Plast Surg. 2007 Sep-Oct;31(5):501-5. doi: 10.1007/s00266-006-0136-2. Epub 2007 Jul 25. PMID 17653684
- [Background] Hu S, Zhang H, Feng Y, Yang Y, Han X, Han X, Zhong Y, Shi J. Introduction of an easy technique for purification and injection of autogenous free fat parcels in correcting of facial contour deformities. Ann Plast Surg. 2007 Jun;58(6):602-7. doi: 10.1097/01.sap.0000248110.59452.49. PMID 17522480
- [Background] Kaufman MR, Bradley JP, Dickinson B, Heller JB, Wasson K, O'Hara C, Huang C, Gabbay J, Ghadjar K, Miller TA. Autologous fat transfer national consensus survey: trends in techniques for harvest, preparation, and application, and perception of short- and long-term results. Plast Reconstr Surg. 2007 Jan;119(1):323-331. doi: 10.1097/01.prs.0000244903.51440.8c. PMID 17255689
- [Background] Sardesai MG, Moore CC. Quantitative and qualitative dermal change with microfat grafting of facial scars. Otolaryngol Head Neck Surg. 2007 Dec;137(6):868-72. doi: 10.1016/j.otohns.2007.08.008. PMID 18036412
- [Background] Coleman SR. Structural fat grafting: more than a permanent filler. Plast Reconstr Surg. 2006 Sep;118(3 Suppl):108S-120S. doi: 10.1097/01.prs.0000234610.81672.e7. PMID 16936550
- [Background] Domergue S, Psomas C, Yachouh J, Lesnik A, Reynes J, Goudot P, Jammet P. Fat microinfiltration autografting for facial restructuring in HIV patients. J Craniomaxillofac Surg. 2006 Dec;34(8):484-8. doi: 10.1016/j.jcms.2006.07.857. Epub 2006 Dec 8. PMID 17157518
- [Background] Narins RS, Tope WD, Pope K, Ross EV. Overtreatment effects associated with a radiofrequency tissue-tightening device: rare, preventable, and correctable with subcision and autologous fat transfer. Dermatol Surg. 2006 Jan;32(1):115-24. doi: 10.1111/1524-4725.2006.32019. No abstract available. PMID 16393612
- [Background] Pontius AT, Williams EF 3rd. The evolution of midface rejuvenation: combining the midface-lift and fat transfer. Arch Facial Plast Surg. 2006 Sep-Oct;8(5):300-5. doi: 10.1001/archfaci.8.5.300. PMID 16982984
- [Background] Burnouf M, Buffet M, Schwarzinger M, Roman P, Bui P, Prevot M, Deleuze J, Morini JP, Franck N, Gorin I, Dupin N. Evaluation of Coleman lipostructure for treatment of facial lipoatrophy in patients with human immunodeficiency virus and parameters associated with the efficiency of this technique. Arch Dermatol. 2005 Oct;141(10):1220-4. doi: 10.1001/archderm.141.10.1220. PMID 16230558
- [Background] Ellenbogen R, Motykie G, Youn A, Svehlak S, Yamini D. Facial reshaping using less invasive methods. Aesthet Surg J. 2005 Mar-Apr;25(2):144-52. doi: 10.1016/j.asj.2005.02.001. PMID 19338805
- [Background] Guaraldi G, Orlando G, De Fazio D, De Lorenzi I, Rottino A, De Santis G, Pedone A, Spaggiari A, Baccarani A, Borghi V, Esposito R. Comparison of three different interventions for the correction of HIV-associated facial lipoatrophy: a prospective study. Antivir Ther. 2005;10(6):753-9. PMID 16218175
- [Background] Kanchwala SK, Holloway L, Bucky LP. Reliable soft tissue augmentation: a clinical comparison of injectable soft-tissue fillers for facial-volume augmentation. Ann Plast Surg. 2005 Jul;55(1):30-5; discussion 35. doi: 10.1097/01.sap.0000168292.69753.73. PMID 15985788
- [Background] Kuran I, Tumerdem B. A new simple method used to prepare fat for injection. Aesthetic Plast Surg. 2005 Jan-Feb;29(1):18-22; discussion 23. doi: 10.1007/s00266-004-0059-8. Epub 2005 Mar 10. PMID 15759091
- [Background] Ellenbogen R, Youn A, Yamini D, Svehlak S. The volumetric face lift. Aesthet Surg J. 2004 Nov-Dec;24(6):514-22. doi: 10.1016/j.asj.2004.08.006. PMID 19336203
- [Background] Karabulut AB, Tumerdem B. Obtaining predictable results in malar augmentation with preimplant fat injection. Plast Reconstr Surg. 2004 Dec;114(7):1974-5. doi: 10.1097/01.prs.0000143917.52057.2a. No abstract available. PMID 15577385
- [Background] Serra-Renom JM, Fontdevila J. Treatment of facial fat atrophy related to treatment with protease inhibitors by autologous fat injection in patients with human immunodeficiency virus infection. Plast Reconstr Surg. 2004 Aug;114(2):551-5; discussion 556-7. doi: 10.1097/01.prs.0000128427.54445.63. PMID 15277830
- [Background] Dasiou-Plakida D. Fat injections for facial rejuvenation: 17 years experience in 1720 patients. J Cosmet Dermatol. 2003 Jul;2(3-4):119-25. doi: 10.1111/j.1473-2130.2004.00060.x. PMID 17163916
- [Background] Sadick NS, Hudgins LC. Fatty acid analysis of transplanted adipose tissue. Arch Dermatol. 2001 Jun;137(6):723-7. PMID 11405760
- [Background] Berman M. Rejuvenation of the upper eyelid complex with autologous fat transplantation. Dermatol Surg. 2000 Dec;26(12):1113-6. PMID 11134987
- [Background] Cortese A, Savastano G, Felicetta L. Free fat transplantation for facial tissue augmentation. J Oral Maxillofac Surg. 2000 Feb;58(2):164-9; discussion 169-70. doi: 10.1016/s0278-2391(00)90331-8. PMID 10670595
- [Background] Erol OO. Facial autologous soft-tissue contouring by adjunction of tissue cocktail injection (micrograft and minigraft mixture of dermis, fascia, and fat). Plast Reconstr Surg. 2000 Nov;106(6):1375-87; discussion 1388-9. doi: 10.1097/00006534-200011000-00026. PMID 11083572
- [Background] Reiche-Fischel O, Wolford LM, Pitta M. Facial contour reconstruction using an autologous free fat graft: a case report with 18-year follow-up. J Oral Maxillofac Surg. 2000 Jan;58(1):103-6. doi: 10.1016/s0278-2391(00)80026-9. No abstract available. PMID 10632174
- [Background] Guerrerosantos J. Simultaneous rhytidoplasty and lipoinjection: a comprehensive aesthetic surgical strategy. Plast Reconstr Surg. 1998 Jul;102(1):191-9. doi: 10.1097/00006534-199807000-00032. PMID 9655427
- [Background] Robinson E, Rumsey N, Partridge J. An evaluation of the impact of social interaction skills training for facially disfigured people. Br J Plast Surg. 1996 Jul;49(5):281-9. doi: 10.1016/s0007-1226(96)90156-3. PMID 8774241
- [Background] Sarwer DB, Crerand CE. Body image and cosmetic medical treatments. Body Image. 2004 Jan;1(1):99-111. doi: 10.1016/S1740-1445(03)00003-2. PMID 18089144
- [Background] Perry S, Difede J, Musngi G, Frances AJ, Jacobsberg L. Predictors of posttraumatic stress disorder after burn injury. Am J Psychiatry. 1992 Jul;149(7):931-5. doi: 10.1176/ajp.149.7.931. PMID 1609874
- [Background] Valente SM. Visual disfigurement and depression. Plast Surg Nurs. 2009 Jan-Mar;29(1):10-6; quiz 17-8. doi: 10.1097/01.PSN.0000347718.75285.23. PMID 19289942
- [Background] Levine E, Degutis L, Pruzinsky T, Shin J, Persing JA. Quality of life and facial trauma: psychological and body image effects. Ann Plast Surg. 2005 May;54(5):502-10. doi: 10.1097/01.sap.0000155282.48465.94. PMID 15838211
- [Background] Guyuron B, Majzoub RK. Facial augmentation with core fat graft: a preliminary report. Plast Reconstr Surg. 2007 Jul;120(1):295-302. doi: 10.1097/01.prs.0000264399.40701.71. PMID 17572578
- [Background] Bisson JI, Shepherd JP, Dhutia M. Psychological sequelae of facial trauma. J Trauma. 1997 Sep;43(3):496-500. doi: 10.1097/00005373-199709000-00018. PMID 9314314
- [Background] Balakrishnan C, Hashim M, Gao D. The effect of partial-thickness facial burns on social functioning. J Burn Care Rehabil. 1999 May-Jun;20(3):224-5. doi: 10.1097/00004630-199905000-00012. PMID 10342476
- [Background] Macgregor FC. Facial disfigurement: problems and management of social interaction and implications for mental health. Aesthetic Plast Surg. 1990 Fall;14(4):249-57. doi: 10.1007/BF01578358. PMID 2239515
- [Background] Thompson A, Kent G. Adjusting to disfigurement: processes involved in dealing with being visibly different. Clin Psychol Rev. 2001 Jul;21(5):663-82. doi: 10.1016/s0272-7358(00)00056-8. PMID 11434225
- [Background] Wallis H, Renneberg B, Ripper S, Germann G, Wind G, Jester A. Emotional distress and psychosocial resources in patients recovering from severe burn injury. J Burn Care Res. 2006 Sep-Oct;27(5):734-41. doi: 10.1097/01.BCR.0000238094.33426.0D. PMID 16998408
- [Background] Yee A, Adjei N, Do J, Ford M, Finkelstein J. Do patient expectations of spinal surgery relate to functional outcome? Clin Orthop Relat Res. 2008 May;466(5):1154-61. doi: 10.1007/s11999-008-0194-7. Epub 2008 Mar 18. PMID 18347892
- [Background] Nguyen TD, Attkisson CC, Stegner BL. Assessment of patient satisfaction: development and refinement of a service evaluation questionnaire. Eval Program Plann. 1983;6(3-4):299-313. doi: 10.1016/0149-7189(83)90010-1. PMID 10267258
- [Background] Weissman MM, Bothwell S. Assessment of social adjustment by patient self-report. Arch Gen Psychiatry. 1976 Sep;33(9):1111-5. doi: 10.1001/archpsyc.1976.01770090101010. PMID 962494
- [Background] Watson D, Friend R. Measurement of social-evaluative anxiety. J Consult Clin Psychol. 1969 Aug;33(4):448-57. doi: 10.1037/h0027806. No abstract available. PMID 5810590
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Weathers FW, Litz BT, Herman DS, Huska JA, Keane TM. The PTSD Checklist: Reliability, validity and diagnostic utility. Paper presented at the Annual Meeting of the International Society for Traumatic Stress Studies; 1993, San Antonio, TX.
- [Background] Rosenberg, M. (1979). Conceiving the self. NY: Basic Books
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Carver CS, Scheier MF, Weintraub JK. Assessing coping strategies: a theoretically based approach. J Pers Soc Psychol. 1989 Feb;56(2):267-83. doi: 10.1037//0022-3514.56.2.267. PMID 2926629
- [Background] Procidano ME, Heller K. Measures of perceived social support from friends and from family: three validation studies. Am J Community Psychol. 1983 Feb;11(1):1-24. doi: 10.1007/BF00898416. PMID 6837532
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Ware J, Kosinski M, Keller S. SF-36 Physical and mental heatlh summary scales: A users manual. 2nd ed. Boston: New England Medical Center, 1994
- [Background] Lawrence J, Heinberg LJ, Roca A, Munster AM, Fauerbach JA. Development and validation of the Satisfaction with Appearance Scale: assessing body image among burn-injured patients. Psychological Assessment 1998; 10: 64-70.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment will come from subjects who have successfully completed IRB# PRO09060101 entitled "Structural Fat Grafting for Craniofacial Trauma". These subjects have expressed a strong desire to participate in this study and have been asked to sign the Research Registry IRB#PRO07050333.
Groups:
- Repeat Facial Fat Grafting: Repeat Fat grafting: treat 5 subjects from protocol IRB # PRO09060101 with an additional fat graft treatment to assess whether this will increase fat graft retention over time.
Period: Overall Study
Arm/Group | Repeat Facial Fat Grafting
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Repeat Facial Fat Grafting: Repeat Fat grafting: Fat grafting is a minimally invasive clinical procedure that has been widely used by plastic surgeons within reconstructive surgery for many years. We treat 5 subjects from protocol (IRB # PRO09060101) with an additional fat graft treatment to assess whether this will increase fat graft retention over time. .
Arm/Group | Repeat Facial Fat Grafting
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants] — 18 years or older
  Participants
    <=18 years | 0
    Between 18 and 65 years | 5
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5
Serial computer tomography imaging [Count of Participants; unit: Participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Facial Volume Score
Description: the facial volume and appearance grading scale evaluates each aesthetic region in the face based on both physical examination and 3D photography by the clinician. scale ranges from 1-3 where a score of 1 indicates an obvious contour defect; 2 shows a noticeable improvement in contour but not sufficient to impart a normal appearance; 3 represents a normal appearance and/or close approximation with a normal uninjured contralateral structure.
Time Frame: assessed at baseline (pre-op), days 7-21 post-op, 3 months post-op, and 9 months post-op
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Facial Volume Score at Baseline: facial volume score at baseline, pre-op
- Facial Volume Score at 7-21 Day PO: facial volume score at 7-21 days post-operation
- Facial Volume Score at 3 Month PO; Facial Volume Score at 9 Months PO: facial volume score at 3 months post-operation
Arm/Group | Facial Volume Score at Baseline | Facial Volume Score at 7-21 Day PO | Facial Volume Score at 3 Month PO | Facial Volume Score at 9 Months PO
Number analyzed (Participants) | 5 | 5 | 5 | 5
units on a scale | 1.8 (0.4) | 2.2 (0.5) | 2.2 (0.4) | 2.6 (0.5)

2. Secondary Outcome: Serial Computed Tomography Imaging
Description: serial computed tomography images were collected to evaluate the volume of the defect
Time Frame: assessed at 7-21 days, 3 months and 9 months post op.
Measure: Mean (Standard Deviation); unit: volume, mL
Groups:
- CT Imaging at 7-21 Days PO: CT imaging at 7-21 days post-operation
- CT Imaging at 3 Months PO: CT imaging at 3 months post-operation
- CT Imaging at 9 Months PO: CT imaging at 9 months post-operation
Arm/Group | CT Imaging at 7-21 Days PO | CT Imaging at 3 Months PO | CT Imaging at 9 Months PO
Number analyzed (Participants) | 3 | 3 | 1
volume, mL | 15 (12.3) | 10.3 (9.1) | 12.4 (NA) — one participant analyzed

ADVERSE EVENTS:
Arm/Group | Repeat Facial Fat Grafting
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Repeat Facial Fat Grafting (N=5)
bruising (Surgical and medical procedures) | 5 (5)
swelling (Surgical and medical procedures) | 5 (5)
pain (Surgical and medical procedures) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes